CLINICAL TRIAL: NCT06877884
Title: A Prospective Registry for Collecting Standardized, Routine Care Data to Characterize Patients, Treatment Patterns, Safety and Treatment Effectiveness in Adult Oncology Patients
Brief Title: A Prospective Registry to Enable Collection of Standardized Routine Care Oncology Patient Data
Status: Recruiting | Type: Observational
Sponsor: N-Power Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: NPM-001
Record Dates: First submitted 2025-02-11; First posted 2025-03-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational registry for patients at participating oncology centers. The data collection includes but is not limited to baseline variables, treatments given and outcome data. Patient surveys are also included. The aim of the study is to generate rich and standardized data for patients and to help enable more patients participate in clinical trials and contribute to research and development.

DETAILED DESCRIPTION:
This is an observational registry for patients at participating oncology centers. The data collection includes but is not limited to baseline variables, treatments given and outcome data. Patient surveys are also included. The aim of the study is to generate rich and standardized data for patients and to help enable more patients participate in clinical trials and contribute to research and development.

ELIGIBILITY:
Inclusion Criteria:

Be a patient at a site (oncology) participating in the Registry Be at least 18 years old Be able and willing to provide signed informed consent

Exclusion Criteria:

Prisoners/imprisonment at time of screening for eligibility Patients who cannot consent without utilization of a legally authorized representative

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients at oncology sites participating in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Effectiveness - Time to treatment discontinuation | This is an open-ended registry where data will be collected, analysed and presented regularly over time.
  Effectiveness outcomes of treatments used in routine clinical care (such as for instance time to treatment discontinuation ) will be captured

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Pacific Cancer Care, Monterey, California
  - Bayhealth Cancer Center-Kent, Dover, Delaware
  - Bayhealth Cancer Center- Sussex, Milford, Delaware
  - Northwest Oncology & Hematology, Elk Grove Village, Illinois
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Lankenau Medical Center, Paoli, Pennsylvania
  - Oncology Consultants, P.A., Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided